CLINICAL TRIAL: NCT03408457
Title: Influence of Perioperative Fluid Balance on Serum Concentrations of Antibiotics and Surgical Site Infections
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Dr. Serge Thal, Principal Investigator, Johannes Gutenberg University Mainz
Other Study IDs: 837.402.17 (11236); U1111-1207-8265 (Registry Identifier: UTN)
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Antibiotic; Anti-Bacterial Agents; Surgical Wound Infection
Keywords: Surgical wound infection; antibiotic concentration; blood level
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Blood sampling after antibiotic administration — Sampling of 6 x 8 mL (in sum 48 mL) via the central venous line (established for the surgical procedure) until postoperative day 2

SUMMARY:
This study evaluates antibiotic serum concentrations in correlation with perioperative fluid balance. Patients will be recruited in rectum and esophageal surgery (representative for low blood loss and restrictive fluid management) and in liver surgery (representative for high blood loss and liberal fluid management). The hypothesis is that high blood loss and liberal fluid management dilute antibiotic serum concentrations thereby potentially increasing surgical site infections.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery of rectom, esophagus or liver with indication for a central venous catheter
* informed consent

Exclusion Criteria:

* pregnancy
* medical emergency
* participation in another study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Surgical Patients of the University Medical Center Mainz
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Serum concentration of antibiotic | 2 days
  ug/mL

SECONDARY OUTCOMES:
Surgical wound infection | 30 days
  Incidence

CONTACTS AND LOCATIONS:
Overall Officials: Serge C Thal, MD PhD, Principal Investigator — University Medical Center of the Johannes Gutenberg-University Mainz
Locations (1):
- Medical Center of the Johannes Gutenberg-University Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No